CLINICAL TRIAL: NCT06381544
Title: The Effect of Aromatherapy Use in Nursing Skills Training on Learning and Anxiety Level: Randomized Controlled Study
Brief Title: The Effect of Aromatherapy Use in Nursing Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Hülya Elmali Simsek, Nursing Program coordinator, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: fbu_nurs_elmali_002
Record Dates: First submitted 2024-03-11; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Nursing Students
Keywords: skills training; nursing students; aromatherapy; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): Aromatherapy Group Aromatherapy will be carried out by spreading the essential oil in the laboratory with the help of a censer. For each censer, 6drops of essential oil mixture (oil mixture ratio, lemon, orange, frankincense oils; 2:2:2 ratio) and two censers will be used. Students will fill out the Introductory Information Form and State Anxiety Scale before being admitted to the laboratory. Students in the experimental group will be taken to the laboratory where aromatherapy is applied, intravenous catheter application will be demonstrated on a simulation model by the researcher during skill training, and each student will practice on the model once. At the end of the application, after students fill out the State Anxiety Scale again, they will be taken to a different room/laboratory and evaluated for skill learning.
  Interventions: Other: Aromatherapy application
- Control (No Intervention): No Intervention: Routine practices Students will fill out the Introductory Information Form and State Anxiety Scale before being admitted to the laboratory. First, the students in the control group will be taken to the laboratory, during the skills training, the intravenous catheter application will be demonstrated on a simulation model by the researcher, and each student will practice on the model once. At the end of the application, after students fill out the State Anxiety Scale again, they will be taken to a different room/laboratory and evaluated for skill learning. The evaluation will be carried out by the researchers for each student individually and with a standard check-list.

INTERVENTIONS:
Other: Aromatherapy application — Applying lemon, orange and frankincense oils via inhalation
  Arms: Aromatherapy

SUMMARY:
Nursing education is an education in which theory and practice are intertwined and requires the development of both cognitive and motor skills of students. The laboratory environment is a bridge between classroom learning and clinical practice. In order for students to transform the target behavior into a skill, it takes place in the laboratory on inanimate models under the supervision of the instructor. It has been assumed that there is a strong relationship between learning and anxiety; while a moderate level of anxiety is necessary for learning, a high level of anxiety causes a decrease in learning.

Many studies have reported that students experience anxiety before their first clinical/practice experience. During skills training, it is observed that students are stressed, their hands are shaking, and they do not feel comfortable, especially before practices involving invasive interventions. This is a factor that makes learning skills training difficult. Therefore, it is important for the student to be comfortable, self-confident, and mentally open to learning during skill training. New applications and different techniques for skill training are important in this sense. It is reported that aromatherapy application has positive effects on reducing anxiety and increasing concentration.

RESEARCH HYPOTHESES:

H0: Aromatherapy has no effect on students' anxiety and learning levels during skill training.

H1: Aromatherapy reduces the anxiety experienced by students during skills training.

H2: Aromatherapy has a positive effect on students' learning nursing skills.

DETAILED DESCRIPTION:
The population of the research consists of 81 students enrolled in the first year of nursing. Power analysis was performed to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 program. As a similar study in the relevant literature, the effect size regarding stress change was calculated as 0.760. In order to exceed the 95% value in determining the power of the study; At a significance level of 5% and an effect size of 0.760, 42 people, 21 people in the groups, need to be reached (df=20; t=1.725). To avoid bias in the people to be included in the study, they were recruited by randomization according to the order of arrival. The randomization table was created using "https://www.calculatorsoup.com". In the research, it was reached a total of 77 students (experiment=39, control=38).

Introductory Information Form, State-Trait Anxiety Inventory and IV Catheter Application Check List will be used to collect data.

In this study, it is planned to analyze the data in SPSS program. Normality tests, mean, standard deviation, minimum, maximum, number-percentage distributions in data analysis; Independent Groups t-test, Mann Whitney U test, One-Way Analysis of Variance, Kruskal-Wallis test will be used. Differences between groups in terms of categorical variables will be examined with the chi-square test. Pearson correlation analysis will be used to examine the relationships between variables, and Cohen-d effect size will be used to determine the effect size.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any respiratory system disease (asthma, COPD, etc.),
* Not having a cardiovascular disease,
* Not being allergic to any odor,
* Lack of pregnancy,
* Not having any obstacle to smell,
* Not using any medication that will affect heart rate and blood pressure,
* It is the absence of a psychiatric disease.

Exclusion Criteria:

* Filling out forms incompletely,
* Not agreeing to participate in the study,
* Having previously received skills training for IV catheter application,
* Any side effects occur during application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Difference between skill learning of students in the aromatherapy group and the control group | immediately after intervention
  Determining the effect of aromatherapy application on nursing students' skill scores.

SECONDARY OUTCOMES:
Difference between anxiety levels of students in the aromatherapy group and the control group | immediately after intervention
  Determining the effect of aromatherapy application on the state anxiety scale scores of nursing students.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Fenerbahce University, Istanbul, Atasehir
  - Fenerbahce University, Ataşehir, Istanbul

IPD SHARING:
Plan to Share IPD: No